CLINICAL TRIAL: NCT02475668
Title: SpO2 Accuracy Validation of Pulse Oximetry Systems During Motion and Non-Motion Conditions of Induced Hypoxia as Compared to Arterial Blood CO-Oximetry
Brief Title: SpO2 Accuracy Validation of Pulse Oximetry Systems During Motion and Non-Motion Conditions
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: QATP2759
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse oximeter — Hypoxia

SUMMARY:
Study to evaluate the %SpO2 accuracy performance of the Nonin Medical pulse oximetry systems.

DETAILED DESCRIPTION:
Study to evaluate the %SpO2 accuracy performance of the Nonin Medical pulse oximetry systems during motion and non-motion.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female
* The subject is of any racial or ethnic group
* The subject is > 30 kg (>66 pounds) in weight (self-reported)
* The subject has at least one finger height of 0.2 - 1.0 inch (based on measurement)
* The subject is between 18 years and 45 years of age (self=reported)
* The subject shows no evidence of medical problems as indicated by satisfactory completion of the health assessment form
* The subject has given written informed consent to participate in the study
* The subject is both willing and able to comply with study procedures.

Exclusion Criteria:

* The subject has a BMI greater than 31 (based on weight and height)
* The subject has had any relevant injury at the sensor location site (self-reported)
* The subject has deformities or abnormalities that may prevent proper application of the device under test (based on examination)
* The subject is current smoker (self-reported)
* The subject has a known respiratory condition (self-reported)
* The subject has a known heart or cardiovascular condition (self-reported)
* The subject is currently pregnant (self-reported)
* The subject is actively trying to get pregnant (self-reported)
* The subject has a clotting disorder (self-reported)
* The subject has Raynaud's Disease (self-reported)
* The subject is known to have a hemoglobinopathy (self-reported)
* The subject is on blood thinners or medication with aspirin (self-reported)
* The subject has unacceptable collateral circulation from the ulnar artery (based on examination)
* The subject is unwilling or unable to provide written informed consent to participate in the study
* The subject is unwilling or unable to comply with the study procedures
* The subject has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
accuracy value (Arms) for %SpO2 over the range of 70-100% in motion and non-motion | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Dave Ransom, MD, Principal Investigator — Avista Adventis Hospital
Locations (1):
- Clinimark, Louisville, Colorado, United States